CLINICAL TRIAL: NCT03267264
Title: Nucleus Claims Study: Evaluating the User Performance and Experience of Nucleus Pen vs. Commercially Available Pen Needle
Brief Title: Evaluating the User Performance and Experience of Nucleus Pen vs. Commercially Available Pen Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DBC-17NUCL07
Record Dates: First submitted 2017-08-22; First posted 2017-08-30 (Actual); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Group 1 (Experimental)
  Interventions: Device: BD Nano™ vs Nucleus
- Group 2 (Experimental)
  Interventions: Device: NovoFine® vs Nucleus
- Group 3 (Experimental)
  Interventions: Device: NovoTwist®/NovoFine® Plus vs Nucleus
- Group 4 (Experimental)
  Interventions: Device: Other Commercially Available Pen Needles (Unifine® Pentips®/Mylife Clickfine®) vs Nucleus

INTERVENTIONS:
Device: BD Nano™ vs Nucleus — Subjects will be randomized to
  1. Nucleus pen needle for the first 15-day period, or current pen needle (BD Nano™) for the second 15-day period or
  2. subject's current pen needle (BD Nano™) for the first 15-day period, Nucleus pen needle for the second 15-day period
  Arms: Group 1
Device: NovoFine® vs Nucleus — Subjects will be randomized to
  1. Nucleus pen needle for the first 15-day period, or current pen needle (NovoFine®) for the second 15-day period or
  2. subject's current pen needle (NovoFine®) for the first 15-day period, Nucleus pen needle for the second 15-day period
  Arms: Group 2
Device: NovoTwist®/NovoFine® Plus vs Nucleus — Subjects will be randomized to
  1. Nucleus pen needle for the first 15-day period, or current pen needle (NovoTwist®/NovoFine Plus®) for the second 15-day period or
  2. subject's current pen needle (NovoTwis®t/NovoFine® Plus) for the first 15-day period, Nucleus pen needle for the second 15-day period
  Arms: Group 3
Device: Other Commercially Available Pen Needles (Unifine® Pentips®/Mylife Clickfine®) vs Nucleus — Subjects will be randomized to
  1. Nucleus pen needle for the first 15-day period, or current pen needle (Other Commercially Available Pen Needles) for the second 15-day period or
  2. subject's current pen needle (Other Commercially Available Pen Needles) for the first 15-day period, Nucleus pen needle for the second 15-day period
  Arms: Group 4

SUMMARY:
This is a multi-site, prospective, open-label, randomized, 2 period cross over study comparing the subjects' current 32G pen needle (four groups of pen needles) to the BD Nucleus pen needle. The study will consist of two 15 day periods ( in which the subject will use each pen needle [BD Nucleus pen needle or subject's current pen needle, order randomized] for injection. At the end of the last study period, each subject will be asked to evaluate his or her perceptions using a 150mm relative VAS scale.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 - 75 inclusive)
2. Diagnosed Type 1 or Type 2 diabetes
3. Every effort will be made to recruit approximately 25% Type 1 patients (of the total population, not of each subgroup) (minimum: 10%, maximum: 50%)
4. Every effort will be made to recruit a minimum of 30 subjects with Asian ethnicity (of the total population, not of each subgroup). Ideally, 60 Asian subjects are needed for the study
5. Minimum within the last 4 months experience self-injecting insulin with a pen injector
6. Minimum within the last 2 months experience self-injecting consistently with one of the following available pen needles OR a subject may be enrolled that is using a 31G/32G pen needle that is not longer than 6mm in length who is willing to transfer to one of the following 32G pen needle with a 14 day wash-in period:

   * BD Nano™ 32Gx4mm
   * NovoFine® 32Gx6mm
   * NovoTwist® 32Gx5mm or
   * NovoFine® Plus 32Gx4mm
   * Owen Mumford PenTips 32Gx4mm or
   * Perrigo / Ypsomed ClickFine 32Gx4mm or
   * Other 32G such as UltiMed, MHC, or other private label.
7. Able and willing to provide informed consent/participant form
8. Able and willing to complete all study procedures

Exclusion Criteria:

1. Self-injecting insulin with a pen injector for less than 3 months
2. Planned changes in insulin regimen (increasing or decreasing number of injections per day).
3. Positive pregnancy test (urine)
4. Currently taking anti-platelet therapy or anticoagulants (Use of up to 81 mg per day of aspirin is permitted).
5. History of a bleeding disorder or easy bruising
6. Blood borne infection(s)
7. History of recurrent dermatological conditions or skin disorder (e.g., psoriasis, eczema)
8. Gross skin anomalies and abnormalities (e.g., scars, stretch marks, discolorations, tattoos, superficial masses, acne, inflammation) located at or very close to the injection sites
9. Fear of needles, history of symptomatic low blood pressure or history of fainting (syncope) during hypodermic injections.
10. Use of any prescription analgesic medications within 24 hours of first study injection, and during the study.
11. A current or previous medical or physical condition that, in the opinion of the investigator, would place the patient at risk or make them unable to perform study procedures or has the potential to confound interpretation of the study results.
12. Currently participating in another study
13. Employed by, or currently serving as a contractor or consultant to BD or any insulin, insulin pen, or insulin pen needle manufacturer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - East West Medical Research Institute, Honolulu, Hawaii
  - PMG Research of Raleigh, Raleigh, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Corporation Lane Internal Medicine and Research Center, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whooley S, Briskin T, Gibney M, Blank L, Berube J, Pflug B. Evaluation the User Performance and Experience of a New Pen Needle with Advanced Hub Face Geometry. Poster presented at: American Association of Diabetes Education Annual Conference; 2018 Aug 17-20; Baltimore, MD.
- [Derived] Whooley S, Briskin T, Gibney MA, Blank LR, Berube J, Pflug BK. Evaluating the User Performance and Experience with a Re-Engineered 4 mm x 32G Pen Needle: A Randomized Trial with Similar Length/Gauge Needles. Diabetes Ther. 2019 Apr;10(2):697-712. doi: 10.1007/s13300-019-0585-7. Epub 2019 Feb 27. PMID 30809762

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 4: Other Commercially Available Pen Needles (MHC Easy Touch, Simple Diagnostics Comfor EZ) vs Nucleus: Subjects will be randomized to
  1. Nucleus pen needle for the first 15-day period, or current pen needle (Other Commercially Available Pen Needles) for the second 15-day period or
  2. subject's current pen needle (Other Commercially Available Pen Needles) for the first 15-day period, Nucleus pen needle for the second 15-day period
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 66 | 49 | 68 | 65
Sequence A(Nucleus) | 34 | 25 | 33 | 33
Sequence B(Comparator) | 32 | 24 | 33 | 32
Completed | 65 | 49 | 66 | 61
Not Completed | 1 | 0 | 2 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Group 3: NovoTwist®/NovoFine® Plus vs Nucleus: Subjects will be randomized to
  1. Nucleus pen needle for the first 15-day period, or current pen needle (NovoTwist®/NovoFine Plus®) for the second 15-day period or
  2. subject's current pen needle (NovoTwist®/NovoFine® Plus) for the first 15-day period, Nucleus pen needle for the second 15-day period
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 66 | 49 | 68 | 65 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (13.3) | 56.6 (12.8) | 55.4 (12.2) | 55.2 (11.2) | 55.6 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 25 | 36 | 33 | 128
  Male | 32 | 24 | 32 | 32 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 3 | 1 | 11
  Not Hispanic or Latino | 63 | 45 | 65 | 64 | 237
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 10 | 10 | 13 | 9 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 0 | 2
  Black or African American | 23 | 15 | 15 | 23 | 76
  White | 26 | 17 | 32 | 28 | 103
  More than one race | 6 | 6 | 7 | 5 | 24
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall User Preference -Combined Groups
Description: This is a combined endpoint for all study subjects. User preference is assessed through a single question reported on a 150mm relative VAS scale with the Nucleus Pen labeled at +75 mm and the subject's current pen needle labeled at -75mm. On this scale, zero represents no preference to either pen needle. Relative VAS scores range from -75mm to 75mm; positive scores reflect preference for BD Nucleus and negative scores reflect preference for the comparator (current pen needle).
Time Frame: 30 Days
Population: Per-protocol population; note that one VAS data point was missing.
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- Combined Groups: Nucleus vs all groups combined
Arm/Group | Combined Groups
Number analyzed (Participants) | 225
mm | 17.5 [10.3 to 24.7]
Statistical Analysis 1: Comparison: Combined Groups; Test type: Non-Inferiority — Two-sided 95% confidence intervals is calculated for the average relative rating. A linear model was used to evaluate the pen needle group effect on the response to test whether the groups can be combined (a p-value < 0.05 for the pen needle group effect indicates non-poolability) and to adjust for the order effect. The order of the pen needles used and the group to which the subject belongs were used as covariates. If the lower bound of the CI is > -10mm, we can conclude in non-inferiority; Overall Mean = 17.5, 95% CI 2-sided [10.3 to 24.7]

2. Secondary Outcome: Overall User Preference - Each Comparator Group
Description: This endpoint analyzes data for individual groups. User preference is assessed through a single question reported on a 150mm relative VAS scale with the Nucleus Pen labeled at +75 mm and the subject's current pen needle labeled at -75mm. On this scale, zero represents no preference to either pen needle. Relative VAS scores range from -75mm to 75mm; positive scores reflect preference for BD Nucleus and negative scores reflect preference for the comparator (current pen needle).
Time Frame: 30 Days
Population: Per-protocol population; note that one VAS data point was missing
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- Group 1: BD Nano™ vs Nucleus
- Group 2: NovoFine® vs Nucleus
- Group 3: NovoTwist®/NovoFine® Plus vs Nucleus
- Group 4: Other Commercially Available Pen Needles
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 60 | 42 | 64 | 59
mm | 30.5 [16.8 to 44.3] | 20.6 [4.1 to 37.1] | 6.2 [-7.2 to 19.5] | 12.8 [-1.1 to 26.7]
Statistical Analysis 1: Comparison: Group 1; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 30.5, 95% CI 2-sided [16.8 to 44.3]
Statistical Analysis 2: Comparison: Group 2; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall = 20.6, 95% CI 2-sided [4.1 to 37.1]
Statistical Analysis 3: Comparison: Group 3; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; overal mean = 6.2, 95% CI 2-sided [-7.2 to 19.5]
Statistical Analysis 4: Comparison: Group 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 12.8, 95% CI 2-sided [-1.1 to 26.7]

3. Secondary Outcome: User Experience - All Study Groups Combined
Description: This is a combined endpoint for all study subjects. User experience is assessed through a series of questions reported on a 150mm relative VAS scale with the Nucleus Pen labeled at +75 mm and the subject's current pen needle labeled at -75mm. On this scale, zero represents no preference to either pen needle. Relative VAS scores range from -75mm to 75mm; positive scores reflect preference for BD Nucleus and negative scores reflect preference for the comparator (current pen needle). Questions include the subject's perception of: Overall Comfort, Anxiety Associated with a Needle Stick Injury, Injection Pain, and Ease of Use.
Time Frame: 30 Days
Population: Per-protocol population
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- All Groups Combined: Resutls from comparator pen needle groups combined and compared to NUCLEUS
Arm/Group | All Groups Combined
Number analyzed (Participants) | 226
mm
  Overall Comfort | 18.0 [11.3 to 24.7]
  Anxiety Associated with a Needle Stick Injury | 15.9 [9.9 to 21.8]
  Injection Pain | 15.5 [8.9 to 22.1]
  Ease of Use | 19.7 [13.8 to 25.7]
Statistical Analysis 1: Comparison: All Groups Combined; Overall Comfort; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall mean = 18.0, 95% CI 2-sided [11.3 to 24.7]
Statistical Analysis 2: Comparison: All Groups Combined; Anxiety Associated with a Needle Stick Injury; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 15.9, 95% CI 2-sided [9.9 to 21.8]
Statistical Analysis 3: Comparison: All Groups Combined; Injection Pain; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 15.5, 95% CI 2-sided [8.9 to 22.1]
Statistical Analysis 4: Comparison: All Groups Combined; Ease of Use; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 19.7, 95% CI 2-sided [13.8 to 25.7]

4. Secondary Outcome: User Experience - Each Individual Study Group
Description: This endpoint analyzes data for individual groups. User experience is assessed through a series of questions reported on a 150mm relative VAS scale with the Nucleus Pen labeled at +75 mm and the subject's current pen needle labeled at -75mm. On this scale, zero represents no preference to either pen needle. Relative VAS scores range from -75mm to 75mm; positive scores reflect preference for BD Nucleus and negative scores reflect preference for the comparator (current pen needle). Questions include the subject's perception of: Overall Comfort, Anxiety Associated with a Needle Stick Injury, Injection Pain, and Ease of Use.
Time Frame: 30 Days
Population: Per-protocol population
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 60 | 43 | 64 | 59
mm
  Overall Comfort | 27.8 [14.9 to 40.7] | 20.7 [5.3 to 36.1] | 8.4 [-4 to 20.9] | 15.1 [2.1 to 28.1]
  Anxiety Associated with a Needle Stick Injury | 20.2 [8.9 to 31.6] | 19.4 [6 to 32.8] | 12.9 [1.9 to 23.8] | 11.0 [-0.5 to 22.4]
  Injection Pain | 16.1 [3.4 to 28.8] | 18.6 [3.6 to 33.7] | 7.0 [-5.3 to 19.4] | 20.2 [7.4 to 33.1]
  Ease of Use | 30.7 [19.3 to 42.1] | 18.4 [4.9 to 31.9] | 17.7 [6.7 to 28.8] | 12.0 [0.5 to 23.5]
Statistical Analysis 1: Comparison: Group 1; Overall Comfort; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 27.8, 95% CI 2-sided [14.9 to 40.7]
Statistical Analysis 2: Comparison: Group 1; Anxiety Associated with a needle stick injury; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 20.2, 95% CI 2-sided [8.9 to 31.6]
Statistical Analysis 3: Comparison: Group 1; Injection Pain; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 16.1, 95% CI 2-sided [3.4 to 28.8]
Statistical Analysis 4: Comparison: Group 1; Ease of Use; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 30.7, 95% CI 2-sided [19.3 to 42.1]
Statistical Analysis 5: Comparison: Group 2; Overall Comfort; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 20.7, 95% CI 2-sided [5.3 to 36.1]
Statistical Analysis 6: Comparison: Group 2; Anxiety Associated with a needle stick; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 19.4, 95% CI 2-sided [6 to 32.8]
Statistical Analysis 7: Comparison: Group 2; Injection Pain; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 18.6, 95% CI 2-sided [3.6 to 33.7]
Statistical Analysis 8: Comparison: Group 2; Ease of Use; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 18.4, 95% CI 2-sided [4.9 to 31.9]
Statistical Analysis 9: Comparison: Group 3; Overall Comfort; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 8.4, 95% CI 2-sided [-4.0 to 20.9]
Statistical Analysis 10: Comparison: Group 3; Anxiety Associated with a Needle stick injury; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 12.9, 95% CI 2-sided [1.9 to 23.8]
Statistical Analysis 11: Comparison: Group 3; Injection Pain; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 7.0, 95% CI 2-sided [-5.3 to 19.4]
Statistical Analysis 12: Comparison: Group 3; Ease of Use; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 17.7, 95% CI 2-sided [6.7 to 28.8]
Statistical Analysis 13: Comparison: Group 4; Overall Comfort; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 15.1, 95% CI 2-sided [2.1 to 28.1]
Statistical Analysis 14: Comparison: Group 4; Anxiety Associated with a Needle Stick Injury; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 11.0, 95% CI 2-sided [-0.5 to 22.4]
Statistical Analysis 15: Comparison: Group 4; Injection Pain; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 20.2, 95% CI 2-sided [7.4 to 33.1]
Statistical Analysis 16: Comparison: Group 4; Eae of Use; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Overall Mean = 12.0, 95% CI 2-sided [0.5 to 23.5]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over 6 week period.
Description: Adverse Events and Serious Adverse Events did not differ from clinicaltrials.gov definitions
Groups:
- Nucleus: This arm contains every subject in the study. Because every subject regardless of group recieved Nucleus
- BD Nano: This arm contains only those subjects that recieve BD Nano, included in results section described in group 1.
- NovoFine®: This arm contains only those subjects that recieved NovoFine®, included in results section described in group 2.
- NovoTwist®/NovoFine®: This arm contains only those subjects that recieved NovoTwist®/NovoFine®, included in results section described in group 3.
- Other Commercially Available Pen Needles (Unifine® Pentips®/M: This arm contains only those subjects that recieved Other Commercial Pen Needles, included in results section described in group 4.
Arm/Group | Nucleus | BD Nano | NovoFine® | NovoTwist®/NovoFine® | Other Commercially Available Pen Needles (Unifine® Pentips®/M
All-Cause Mortality (participants affected / at risk) | 0/241 | 0/65 | 0/49 | 0/66 | 0/61
Serious Adverse Events (participants affected / at risk) | 1/241 | 0/65 | 1/49 | 0/66 | 1/61
Other Adverse Events (participants affected / at risk) | 50/241 | 5/65 | 4/49 | 4/66 | 5/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nucleus (N=241) | BD Nano (N=65) | NovoFine® (N=49) | NovoTwist®/NovoFine® (N=66) | Other Commercially Available Pen Needles (Unifine® Pentips®/M (N=61)
Broken Right Ankle (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Subject broke their ankle
Infection of L Hand Laceration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nucleus (N=241) | BD Nano (N=65) | NovoFine® (N=49) | NovoTwist®/NovoFine® (N=66) | Other Commercially Available Pen Needles (Unifine® Pentips®/M (N=61)
Bleeding (Injury, poisoning and procedural complications) | 21 (21) | 4 (4) | 1 (1) | 2 (2) | 2 (2) — Experience exceeds that normally associated with the procedure, as judged by the Subject
Bruising (Injury, poisoning and procedural complications) | 14 (14) | 1 (1) | 0 (0) | 0 (0) | 2 (2) — Experience exceeds that normally associated with the procedure, as judged by the Subject
Swelling/Pain at injection site (Injury, poisoning and procedural complications) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Experience exceeds that normally associated with the procedure, as judged by the Subject
Hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Abcess under chin (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
L hand Laceration (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Worsening of Type 2 Diabetes (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT03267264/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT03267264/SAP_001.pdf